CLINICAL TRIAL: NCT00684021
Title: Transplantation in Myocardial Infarction Evaluation (TIME) Protocol: A Phase II, Randomized, Controlled, Double-Blind Trial Evaluating the Effect of Timing on the Administration of Bone Marrow Mononuclear Cells (BMMNCs) Versus Placebo in Patients With Acute Myocardial Infarction
Brief Title: Use of Adult Autologous Stem Cells in Treating People Who Have Had a Heart Attack (The TIME Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr Lemuel A Moye III, Professor - School of Public Health, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 579; U01HL087318 (NIH); 1 U01-HL-087318-01 (Project 1)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Left Ventricular Dysfunction
Keywords: Acute Myocardial Infarction; Global Left Ventricular Ejection Fraction; Regional Left Ventricular Ejection Fraction; Left Ventricular Mass; Infarct Size; End Systolic Volume; End Diastolic Volume
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Participants will receive active adult stem cell infusion 3 days after percutaneous coronary intervention (PCI).
  Interventions: Biological: Adult stem cells
- 2 (Active Comparator): Participants will receive active adult stem cell infusion 7 days after PCI.
  Interventions: Biological: Adult stem cells
- 3 (Placebo Comparator): Participants will receive placebo infusion (5% human serum albumin [HSA]) 3 days after PCI.
  Interventions: Biological: Placebo
- 4 (Placebo Comparator): Participants will receive placebo infusion (5% HSA) 7 days after PCI.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Adult stem cells — One time infusion of approximately 150 million total nucleated cells (TNC) in 30 ml of 5% HSA/saline solution
  Other Names: Adult autologous stem cells; Bone marrow mononucleated cells
  Arms: 1; 2
Biological: Placebo — One time infusion of 30 ml of HSA (5%)
  Other Names: HSA
  Arms: 3; 4

SUMMARY:
Heart attacks are a leading cause of death for both men and women in the United States. A heart attack occurs when blood flow to the heart is restricted, commonly due to a blood clot that has formed in one of the coronary arteries. If the clot becomes large enough, blood flow to the heart can be blocked almost completely and the heart muscle in that area can suffer permanent injury or death. Although a percutaneous coronary intervention (PCI) can be used to open up the blocked artery and restore blood flow to the heart muscle, there may be a significant amount of heart tissue that has been irreversibly damaged. Recent studies have shown that adult stem cells from bone marrow may be able to improve heart function after a heart attack. This study will evaluate the safety and effectiveness of using adult stem cells for improving heart function in people who have had a recent heart attack and a PCI.

DETAILED DESCRIPTION:
More than 1 million Americans suffer a heart attack each year, resulting in about a 38% mortality rate. Although current treatments are able to stabilize the condition of the heart, none is able to restore heart function as it was prior to the heart attack. The permanent damage to the heart can lead to more severe problems, such as heart failure and irregular heartbeat, making the discovery of treatments to improve heart function after a heart attack important. Adult stem cells, which are immature cells that can become many different types of cells, may offer a potential means of reversing or preventing permanent damage caused by a heart attack. These specialized cells may have the ability to promote blood vessel growth, prevent cell death, and transform themselves into a number of tissues, including muscle. Recent studies have shown promise in using adult stem cells from bone marrow to reverse damage to the heart muscle caused by a heart attack, but more research is needed to assess the safety and effectiveness of stem cell use and to discover the best time to administer treatment. This study will evaluate the safety and effectiveness of placing adult stem cells into injured heart muscle for improving heart function in people who have had a recent heart attack and a PCI. Additionally, this study will help determine the best time to insert stem cells after a heart attack.

Participation in this study will last 24 months. All participants will first undergo baseline assessments that will include a medical history, a physical exam, an electrocardiogram (ECG), blood draws, an echocardiogram, and a magnetic resonance imaging (MRI) test. Participants will then be assigned randomly to receive stem cells or placebo either 3 or 7 days after their heart attack. The morning of the stem cell or placebo infusion, participants will undergo a blood draw and a bone marrow aspiration procedure of the hip bone to collect the stem cells. Later the same day, either stem cells or placebo will be infused through a catheter and into the damaged area of the heart.

For the first 24 hours following the infusion, participants will be asked to wear a small ECG machine called a Holter monitor. Participants will also be asked to record their temperature twice a day for a month after the infusion. Participants will return for follow-up visits at Months 1, 3, 6, 12, and 24 and will repeat many of the baseline assessments.

ELIGIBILITY:
Inclusion criteria

1. Patients at least 21 years of age
2. Patients with first acute MI with successful primary percutaneous coronary intervention (PCI) in an artery at least 2.5 mm in diameter within 24 hours of onset of symptoms.
3. No contraindications to undergoing cell therapy procedure within three to seven days following AMI and PCI.
4. Hemodynamic stability as defined as no requirement for IABP, inotropic or blood pressure supporting medications.
5. Ejection fraction following reperfusion with PCI <=45% as assessed by echocardiography.
6. Consent to protocol and agree to comply with all follow-up visits and studies.
7. Women of child bearing potential willing to use an active form of birth control.

Exclusion criteria

Patients will be excluded from the study if they meet any of the following conditions:

1. History of sustained ventricular arrhythmias not related to their AMI (evidenced by previous holter monitoring and/or medication history for sustained ventricular arrhythmias in patient's medical chart).
2. Require CABG or PCI due to the presence of residual coronary stenosis >70% luminal obstruction in the non-infarct related vessel (Additional PCI of non-culprit vessels may be performed prior to enrollment).
3. History of any malignancy within the past five years excluding non-melanoma skin cancer or cervical cancer in-situ.
4. History of chronic anemia (hemoglobin (Hb) <9.0 mg/dl).
5. History of thrombocytosis (platelets >500k).
6. History of thrombocytopenia in the absence of recent evidence that platelet counts are normal
7. Known history of elevated INR (PT) or PTT.
8. Life expectancy less than one year.
9. History of untreated alcohol or drug abuse.
10. Currently enrolled in another investigational drug or device trial
11. Previous CABG.
12. Previous MI resulting in LV dysfunction (LVEF <55%)
13. History of stroke or transient ischemic attack (TIA) within the past six months.
14. History of severe valvular heart disease (aortic valve area <1.0 cm2 or >3+ mitral regurgitation).
15. Pregnancy or breast feeding
16. Subjects with a known history of HIV, or has active hepatitis B,active hepatitis C, or active TB
17. Patients with active inflammatory or autoimmune disease on chronic immuno-suppressive therapy.
18. Contraindications to cMRI.
19. Previous radiation to the pelvis with white blood cell count (WBC) and platelet counts below hospital specific normal values.
20. Women child bearing potential not willing to practice an active form of birth control.
21. Chronic liver disease that might interfere with survival or treatment with cell therapy.
22. Chronic renal insufficiency as defined by a creatinine ≥ 2.0 mg/dL or requires chronic dialysis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simari, MD, Study Chair — Cardiovascular Cell Therapy Research Network
Locations (5):
- United States (5):
  - University of Florida-Department of Medicine, Gainesville, Florida
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Traverse JH, Henry TD, Vaughan DE, Ellis SG, Pepine CJ, Willerson JT, Zhao DX, Piller LB, Penn MS, Byrne BJ, Perin EC, Gee AP, Hatzopoulos AK, McKenna DH, Forder JR, Taylor DA, Cogle CR, Olson RE, Jorgenson BC, Sayre SL, Vojvodic RW, Gordon DJ, Skarlatos SI, Moye' LA, Simari RD; Cardiovascular Cell Therapy Research Network (CCTRN). Rationale and design for TIME: A phase II, randomized, double-blind, placebo-controlled pilot trial evaluating the safety and effect of timing of administration of bone marrow mononuclear cells after acute myocardial infarction. Am Heart J. 2009 Sep;158(3):356-63. doi: 10.1016/j.ahj.2009.06.009. Epub 2009 Jul 23. PMID 19699857
- [Background] Gee AP, Richman S, Durett A, McKenna D, Traverse J, Henry T, Fisk D, Pepine C, Bloom J, Willerson J, Prater K, Zhao D, Koc JR, Ellis S, Taylor D, Cogle C, Moye L, Simari R, Skarlatos S. Multicenter cell processing for cardiovascular regenerative medicine applications: the Cardiovascular Cell Therapy Research Network (CCTRN) experience. Cytotherapy. 2010 Sep;12(5):684-91. doi: 10.3109/14653249.2010.487900. PMID 20524773
- [Background] Zierold C, Carlson MA, Obodo UC, Wise E, Piazza VA, Meeks MW, Vojvodic RW, Baraniuk S, Henry TD, Gee AP, Ellis SG, Moye LA, Pepine CJ, Cogle CR, Taylor DA. Developing mechanistic insights into cardiovascular cell therapy: Cardiovascular Cell Therapy Research Network Biorepository Core Laboratory rationale. Am Heart J. 2011 Dec;162(6):973-80. doi: 10.1016/j.ahj.2011.05.024. PMID 22137069
- [Result] Traverse JH, Henry TD, Pepine CJ, Willerson JT, Zhao DX, Ellis SG, Forder JR, Anderson RD, Hatzopoulos AK, Penn MS, Perin EC, Chambers J, Baran KW, Raveendran G, Lambert C, Lerman A, Simon DI, Vaughan DE, Lai D, Gee AP, Taylor DA, Cogle CR, Thomas JD, Olson RE, Bowman S, Francescon J, Geither C, Handberg E, Kappenman C, Westbrook L, Piller LB, Simpson LM, Baraniuk S, Loghin C, Aguilar D, Richman S, Zierold C, Spoon DB, Bettencourt J, Sayre SL, Vojvodic RW, Skarlatos SI, Gordon DJ, Ebert RF, Kwak M, Moye LA, Simari RD; Cardiovascular Cell Therapy Research Network (CCTRN). Effect of the use and timing of bone marrow mononuclear cell delivery on left ventricular function after acute myocardial infarction: the TIME randomized trial. JAMA. 2012 Dec 12;308(22):2380-9. doi: 10.1001/jama.2012.28726. PMID 23129008
- [Derived] Traverse JH, Henry TD, Pepine CJ, Willerson JT, Chugh A, Yang PC, Zhao DXM, Ellis SG, Forder JR, Perin EC, Penn MS, Hatzopoulos AK, Chambers JC, Baran KW, Raveendran G, Gee AP, Taylor DA, Moye L, Ebert RF, Simari RD. TIME Trial: Effect of Timing of Stem Cell Delivery Following ST-Elevation Myocardial Infarction on the Recovery of Global and Regional Left Ventricular Function: Final 2-Year Analysis. Circ Res. 2018 Feb 2;122(3):479-488. doi: 10.1161/CIRCRESAHA.117.311466. Epub 2017 Dec 5. PMID 29208679
- [Derived] Schutt RC, Trachtenberg BH, Cooke JP, Traverse JH, Henry TD, Pepine CJ, Willerson JT, Perin EC, Ellis SG, Zhao DX, Bhatnagar A, Johnstone BH, Lai D, Resende M, Ebert RF, Wu JC, Sayre SL, Orozco A, Zierold C, Simari RD, Moye L, Cogle CR, Taylor DA; Cardiovascular Cell Therapy Research Network (CCTRN). Bone marrow characteristics associated with changes in infarct size after STEMI: a biorepository evaluation from the CCTRN TIME trial. Circ Res. 2015 Jan 2;116(1):99-107. doi: 10.1161/CIRCRESAHA.116.304710. Epub 2014 Nov 18. PMID 25406300
- [Derived] Cogle CR, Wise E, Meacham AM, Zierold C, Traverse JH, Henry TD, Perin EC, Willerson JT, Ellis SG, Carlson M, Zhao DX, Bolli R, Cooke JP, Anwaruddin S, Bhatnagar A, da Graca Cabreira-Hansen M, Grant MB, Lai D, Moye L, Ebert RF, Olson RE, Sayre SL, Schulman IH, Bosse RC, Scott EW, Simari RD, Pepine CJ, Taylor DA; Cardiovascular Cell Therapy Research Network (CCTRN). Detailed analysis of bone marrow from patients with ischemic heart disease and left ventricular dysfunction: BM CD34, CD11b, and clonogenic capacity as biomarkers for clinical outcomes. Circ Res. 2014 Oct 24;115(10):867-74. doi: 10.1161/CIRCRESAHA.115.304353. Epub 2014 Aug 18. PMID 25136078
- [Derived] Traverse JH, Henry TD, Pepine CJ, Willerson JT, Ellis SG. One-year follow-up of intracoronary stem cell delivery on left ventricular function following ST-elevation myocardial infarction. JAMA. 2014 Jan 15;311(3):301-2. doi: 10.1001/jama.2013.282674. No abstract available. PMID 24247415
- [Derived] Traverse JH, Henry TD, Vaughan DE, Ellis SG, Pepine CJ, Willerson JT, Zhao DX, Simpson LM, Penn MS, Byrne BJ, Perin EC, Gee AP, Hatzopoulos AK, McKenna DH, Forder JR, Taylor DA, Cogle CR, Baraniuk S, Olson RE, Jorgenson BC, Sayre SL, Vojvodic RW, Gordon DJ, Skarlatos SI, Moye LA, Simari RD; Cardiovascular Cell Therapy Research Network. LateTIME: a phase-II, randomized, double-blinded, placebo-controlled, pilot trial evaluating the safety and effect of administration of bone marrow mononuclear cells 2 to 3 weeks after acute myocardial infarction. Tex Heart Inst J. 2010;37(4):412-20. PMID 20844613
- See also: Click here for more information on this study at the Cardiovascular Cell Therapy Research Network (CCTRN) — http://www.cctrn.org
- See also: Click here for the National Heart, Lung, and Blood Institute — http://www.nhlbi.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at five Network centers and their associated satellite facilities between July 2008 and November 2011. The main centers are located in Ohio, Texas, Florida, Minnesota, and Tennessee. Study brochures, patient informational DVDs, and clinical trials.gov were among the tools used for recruitment.
Groups:
- Day 3 Stem Cell Arm: Participants will receive active adult stem cell infusion 3 days after percutaneous coronary intervention (PCI).
- Day 3 Placebo Arm: Participants will receive placebo infusion (5% human serum albumin [HSA]) 3 days after PCI.
- Day 7 Stem Cell Arm: Participants will receive active adult stem cell infusion 7 days after PCI.
- Day 7 Placebo Arm: Participants will receive placebo infusion (5% HSA) 7 days after PCI.
Period: Overall Study
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Started | 43 | 24 | 36 | 17
Completed | 41 | 22 | 34 | 15
Not Completed | 2 | 2 | 2 | 2
Not completed — MRI Contraindicated | 1 | 1 | 1 | 0
Not completed — MRI not performed | 0 | 1 | 1 | 2
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm | Total
Number analyzed (Participants) | 43 | 24 | 36 | 17 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.8) | 57.0 (12.4) | 58.2 (11.3) | 57.0 (8.0) | 56.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 2 | 15
  Male | 38 | 21 | 31 | 15 | 105
Region of Enrollment [Number; unit: participants]
  United States | 43 | 24 | 36 | 17 | 120

OUTCOME MEASURES:

1. Primary Outcome: Global Left Ventricular Function
Description: Left ventricular ejection fraction (global) as assessed via cardiac MRI. Values reported represent the change in Global EF from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in Global EF from baseline to six months.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 41 | 22 | 34 | 15
percentage of ejection fraction | 3.5 (11.0) | 4.4 (10.6) | 2.8 (9.7) | 1.7 (8.2)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; Test type: Superiority or Other; p = 0.959, t-test, 2 sided; Stem cell treatment arm combined (Day 3 and Day7); placebo group also combined; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-4.1 to 3.9], Standard Error of Mean 2.0

2. Secondary Outcome: Clincal and Safety Outcomes
Description: Number of events -death, reinfarction, repeat revascularizations (target and nontarget vessels) hospitalizations for heart failure, ICD placements
Time Frame: Measured from baseline to six months.
Population: All randomized patients were followed for clinical outcomes.
Measure: Number; unit: events
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 43 | 24 | 36 | 17
events | 10 | 9 | 6 | 1
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; Clinical and Safety Outcomes including death, reinfarction, repeat revascularization, hospitalization for heart failure and ICD placement. The relative incidences of events are compared between the active and placebo groups.However the paucity of events precluded a reliable time to event analysis; Test type: Superiority or Other; p = 0.93, Fisher Exact; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.42 to 2.23]

3. Secondary Outcome: Left Ventricular Mass
Description: Left ventricular mass (LV mass. Values reported represent the change in LV mass from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in LV mass from baseline to six months.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 40 | 22 | 33 | 13
g | -20.4 (22.8) | -13.2 (30.6) | -16.3 (16.7) | -20.7 (26.9)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; Day 3 Stem Cell Arm and Day 7 Stem Cell Arm were combined and compared to the combination of Day 3 Placebo and Day 7 Placebo arms; Test type: Superiority or Other; p = 0.585, Regression, Linear; Mean Difference (Net) = -2.6, 95% CI 2-sided [-12.2 to 6.9], Standard Error of Mean 4.8

4. Secondary Outcome: End Diastolic Volume Index
Description: Left ventricular end diastolic volume index. Values reported represent the change in LV end diastolic index from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in LV end diastolic index from baseline to six months.
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 41 | 22 | 34 | 15
mL/m2 | 11.4 (18.5) | 11.7 (19.8) | 13.3 (19.5) | 9.7 (16.0)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.831, Regression, Linear; Mean Difference (Net) = 0.8, 95% CI 2-sided [-6.6 to 8.2], Standard Error of Mean 3.7

5. Secondary Outcome: End Systolic Volume Index
Description: Left ventricular end systolic volume index. Values reported represent the change in LV end systolic volume index from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in LV end systolic volume index from baseline to six months.
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 41 | 22 | 34 | 15
mL/m2 | 4.1 (15.0) | 4.1 (16.5) | 6.2 (17.4) | 4.6 (12.8)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.817, Regression, Linear; Mean Difference (Net) = 0.7, 95% CI 2-sided [-5.5 to 7.0], Standard Error of Mean 3.7

6. Secondary Outcome: Infarct Volume
Description: Infarct volume(mL). Values reported represent the change in infarct volume from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in infarct volume from baseline to six months.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 40 | 20 | 32 | 13
mL | -9.7 (18.4) | -7.7 (23.4) | -13.6 (18.8) | -5.3 (29.3)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.272, Regression, Linear; Mean Difference (Net) = -4.7, 95% CI 2-sided [-13.7 to 3.67], Standard Error of Mean 4.27

7. Primary Outcome: Regional Left Ventricular Function (Infarct Zone Wall Motion)
Description: One of two calculated values of regional left ventricular function as assessed via cardiac MRI. The infarct zone is defined as the cMRI segments with the largest 2 signal intensity enhancement measures with gadolinium (using a 17-segment model).Values reported represent the change in wall motion over time in the infarct zone from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included. Values reported represent the change in wall motion over time in the infarct zone from baseline to six months.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 41 | 22 | 34 | 15
mm | 2.1 (5.9) | 2.4 (5.3) | 1.2 (4.9) | 2.8 (4.4)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; Test type: Superiority or Other; p = 0.409, t-test, 2 sided; Stem cell treatment arm combined (Day 3 and Day7); placebo group also combined; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.0 to 1.2], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; Test type: Superiority or Other; p = 0.02, Regression, Linear; Mean Difference (Net) = 100, 95% CI 2-sided [15 to 1000], Standard Error of Mean .01

8. Primary Outcome: Regional Left Ventricular Function (Border Zone Wall Motion)
Description: Two of two calculated values of regional left ventricular function assessed via cardiac MRI. The border zone is defined as those regions adjacent to the infarct zone in which the cMRI signal intensity enhancement were in the 10%-75% range. Values reported represent the change in wall motion over time in the border zone of the infarct from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Values reported represent the change in wall motion over time in the border zone of the infarct from baseline to six months.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Number analyzed (Participants) | 41 | 22 | 34 | 15
mm | 3.5 (9.3) | 4.3 (8.7) | 4.2 (8.3) | 4.4 (7.2)
Statistical Analysis 1: Comparison: Day 3 Stem Cell Arm vs Day 3 Placebo Arm vs Day 7 Stem Cell Arm vs Day 7 Placebo Arm; Test type: Superiority or Other; p = 0.777, t-test, 2 sided; Stem cell treatment arm combined (Day 3 and Day7); placebo group also combined; Mean Difference (Net) = -0.5, 95% CI 2-sided [-3.9 to 2.9], Standard Error of Mean 1.7

ADVERSE EVENTS:
Time Frame: Events reported are from Randomization Date to the 6 month endpoint data collection window (i.e. 210 days post intervention)
Arm/Group | Day 3 Stem Cell Arm | Day 3 Placebo Arm | Day 7 Stem Cell Arm | Day 7 Placebo Arm
Serious Adverse Events (participants affected / at risk) | 17/43 | 6/24 | 11/36 | 2/17
Other Adverse Events (participants affected / at risk) | 10/43 | 6/24 | 13/36 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 3 Stem Cell Arm (N=43) | Day 3 Placebo Arm (N=24) | Day 7 Stem Cell Arm (N=36) | Day 7 Placebo Arm (N=17)
Chest Pain (Cardiac disorders) | 8 (9) | 2 (2) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Heart Failure (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
New/Worsening Thrombus (Cardiac disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 3 Stem Cell Arm (N=43) | Day 3 Placebo Arm (N=24) | Day 7 Stem Cell Arm (N=36) | Day 7 Placebo Arm (N=17)
Groin bruising/bleeding (Cardiac disorders) | 5 (6) | 3 (3) | 4 (6) | 4 (5) — Groin bruising or bleeding at site of catheter insertion
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombus (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
The choice of Day 3 or Day 7 as randomization points while based on the literature were nevertheless somewhat arbitrary. cMR-baseed ejection fractions tended to be high.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes